CLINICAL TRIAL: NCT04129450
Title: Group-based Mindfulness for Patients With Chronic Low Back Pain in the Primary Care Setting
Brief Title: Group-based Mindfulness for Chronic Pain in the Primary Care Setting
Acronym: OPTIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-39165; 4UH3AT010621-02 (NIH)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Back Pain
Keywords: Mindfulness-Based Stress Reduction; Medical group visits; Primary care setting
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Pain Program + Usual PCP Care (Experimental): Participants will undergo 8 weekly 90 minute sessions of Mindfulness-Based Stress Reduction in addition to receiving usual PCP care for chronic lower back pain.
  Interventions: Other: Group medical visits with mindfulness-based stress reduction; Other: Usual PCP care
- Usual PCP Care (Active Comparator): Participants will receive usual PCP care for chronic lower back pain.
  Interventions: Other: Usual PCP care

INTERVENTIONS:
Other: Group medical visits with mindfulness-based stress reduction — Eight weekly 90 minute sessions of mindfulness-based stress reduction in group medical visits
  Arms: Mindfulness Pain Program + Usual PCP Care
Other: Usual PCP care — Usual one on one PCP care for chronic lower back pain

SUMMARY:
The purpose of this pragmatic clinical trial (PCT) research is to determine whether a group-visit approach modeled on Mindfulness-Based Stress Reduction can improve function for persons with chronic low back pain. This will be done by an embedded PCT within the evidence-based "OPTIMUM" (Optimizing Pain Treatment In Medical settings Using Mindfulness) program.

DETAILED DESCRIPTION:
The research will be conducted with three health care system (HCS) sites: Boston Medical Center (BMC), MA, a safety net health system; University of Pittsburgh Medical Center (UPMC), Pittsburgh, PA, a large health system; and Piedmont Health Services, NC, a network of federally funded health centers in partnership with the University of North Carolina (UNC), Chapel Hill.

As per NIH protocol for the funding, the first 12 month (Phase 1) of this PCT will be a pilot to plan and test the group-based mindfulness program for chronic pain program in each of the three sites with 5 participants/site. Once completed the Phase 2 will be conducted to integrate and test the group-based mindfulness program compared to standard of care for patients with chronic low back pain (cLBP) in the primary care setting at each collaborating site.

Eligible consenting participants will be randomized to either: the primary care providers (PCP) usual care group, or the group with both PCP usual care and the 8 weeks mindfulness clinical pain group. Participants will be asked to complete baseline and follow-up surveys about pain, function, pain medicine use, mood and anxiety symptoms, and quality of life. The surveys will take up to an hour to complete.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Chronic low back pain, which is pain that persists for at least 3-months and has resulted in pain on at least half the days in the past 6 months
* A score ≥ 3 on the Pain, Enjoyment of Life and General Activity (PEG)
* Willing and able to provide online or telephone informed consent
* Speak English as the intervention manual is currently written in English

Exclusion Criteria:

* Do not meet the above inclusion criteria
* Red flags- recent (past month) worsening of pain, unexplained fever, unexplained weight loss
* Pregnancy
* Metastatic cancer
* First-degree relatives (parents, siblings, child) of someone who has participated or is participating in the OPTIMUM study
* Members of the same household
* Not a patient at a participating clinic or persons not planning to continue as a patient at a participating clinic for 12 or more months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Morone, MD, MS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller VE, Barnhill J, Greco CM, Castro G, Nguyen TP, Gardiner P, Faurot KR, Gaylord S, Weinberg JM, Thomas HN, Sariahmed K, Morone NE. Prevalence of Chronic Overlapping Pain Conditions in Participants With Chronic Low Back Pain Enrolled in a Pragmatic Trial of Mindfulness-Based Stress Reduction. Eur J Pain. 2025 Oct;29(9):e70119. doi: 10.1002/ejp.70119. PMID 40891220
- [Derived] Barnhill JL, Castro G, Lathren C, Harr E, Roth I, Baez JE, Rodriguez R, Lawrence S, Gardiner P, Greco CM, Thomas HN, Gaylord SA, Dore G, Bengert A, Morone NE. The Hidden Complexity of Virtual Mindfulness-Based Group Medical Visits: Comfort, Challenge, and the Influence of Social Determinants of Health. Glob Adv Integr Med Health. 2025 Mar 27;14:27536130251326938. doi: 10.1177/27536130251326938. eCollection 2025 Jan-Dec. PMID 40162193
- [Derived] Greco CM, Gaylord SA, Faurot K, Weinberg JM, Gardiner P, Roth I, Barnhill JL, Thomas HN, Dhamne SC, Lathren C, Baez JE, Lawrence S, Neogi T, Lasser KE, Castro MG, White AM, Simmons SJ, Ferrao C, Binda DD, Elhadidy N, Eason KM, McTigue KM, Morone NE. The design and methods of the OPTIMUM study: A multisite pragmatic randomized clinical trial of a telehealth group mindfulness program for persons with chronic low back pain. Contemp Clin Trials. 2021 Oct;109:106545. doi: 10.1016/j.cct.2021.106545. Epub 2021 Aug 27. PMID 34455111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Internal Medicine Clinic at Boston Medical Center (BMC), University of Pittsburgh, University of North Carolina (UNC) at Chapel Hill in partnership with Piedmont Health and UNC HealthCare by trained and IRB-approved staff. Ways for recruiting included flyers throughout the clinics, provider referral, automated electronic medical record review, clinic sign-up sheet, and website.
Pre-assignment Details: Of 451 enrolled participants, 224 were assigned to the intervention and 227 to the control group.
Groups:
- Mindfulness Pain Program + Usual Primary Care Provider (PCP) Care: Participants will undergo 8 weekly 90 minute sessions of Mindfulness-Based Stress Reduction in addition to receiving usual Primary Care Provider (PCP) care for chronic lower back pain.
Period: Overall Study
Arm/Group | Mindfulness Pain Program + Usual Primary Care Provider (PCP) Care | Usual PCP Care
Started | 224 | 227
Completed | 190 | 212
Not Completed | 34 | 15
Not completed — Lost to Follow-up | 20 | 10
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Work Family Obligations | 2 | 0
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Pain Program + Usual PCP Care | Usual PCP Care | Total
Number analyzed (Participants) | 224 | 227 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (14.4) | 51.9 (14.95) | 52.13 (14.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Baseline: Female | 156 | 162 | 318
  Baseline: Male | 67 | 65 | 132
  Baseline: Intersex | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Baseline: Non-Hispanic black | 91 | 96 | 187
  Baseline: Non-Hispanic white | 100 | 104 | 204
  Baseline: Hispanic | 13 | 17 | 30
  Baseline: Other | 15 | 9 | 24
  Baseline: Unknown | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 224 | 227 | 451

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity and Interference at Baseline, 8 Weeks, 6 Months (Primary Timepoint), & 12 Months: Pain, Enjoyment, General Activity (PEG) Score
Description: The PEG (pain, enjoyment, general activity) composite score will be used to assess pain intensity and interference. The PEG is a 3 item score with potential responses of 0 to 10 with 10 being the most severe pain. The 3 PEG items referring to the past week are: average pain, how pain interfered with enjoyment of life, how pain interfered with general activity To compute the PEG score, add the responses to the questions above, then divide by three to get a final score out of 10.
Time Frame: Baseline, 8 weeks, 6 months (primary timepoint), 12 months
Population: Persons with chronic low back pain 18 years old or older.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Pain Program + Usual PCP Care | Usual PCP Care
Number analyzed (Participants) | 224 | 227
score on a scale
  Baseline | 6.37 [5.95 to 6.79] | 5.87 [5.45 to 6.29]
  8 weeks | 5.21 [4.76 to 5.65] | 5.6 [5.16 to 6.04]
  6 months | 5.16 [4.69 to 5.62] | 5.28 [4.83 to 5.74]
  12 Months | 4.85 [4.39 to 5.3] | 5.09 [4.65 to 5.54]

2. Secondary Outcome: Physical Function at Baseline, 8 Weeks, 6 Months, and 12 Months
Description: Physical function will be assessed using the 4 items Patient Reported Outcome Measurement Information System (PROMIS) at 8 weeks and 12 months and the 6 items PROMIS assessment at baseline and 6 months. It measures self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back). For the 4 items PROMIS, each question usually has five response options ranging in value from one to five. Raw scores range from 4 to 20, and t-scores range from 22.5 to 57. For the 6 items PROMIS, each question usually has five response options ranging in value from one to five. Raw scores range from 6 to 30, t-scores range from 21 to 59. Higher scores are more favorable.
Time Frame: Baseline, 8 weeks, 6 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

3. Secondary Outcome: Sleep Disturbance at Baseline, 8 Weeks, 6 Months, & 12 Months
Description: Sleep disturbance will be assessed using the 4 items PROMIS at 8 weeks and 12 months and the 6 items PROMIS assessment at baseline and 6 months. It assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. For the 4 items PROMIS, each question usually has five response options ranging in value from one to five. Raw scores range from 4 to 20, and t-scores range from 32 to 73.3. For the 6 items PROMIS, each question usually has five response options ranging in value from one to five. Raw scores range from 6 to 30, t-scores range from 31.7 to 76.1. Higher scores indicate worsen sleep disturbance.
Time Frame: Baseline, 8 weeks, 6 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Quality of Life at Baseline, 8 Weeks, 6 Months, & 12 Months
Description: Quality of life will be assessed using the PROMIS-29+2 Profile v2.1 (PROPr) at baseline, 8 weeks, 6 months, & 12 months. The PROPr assesses pain intensity using a single 0-10 numeric rating item and eight health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, sleep disturbance, and cognitive function abilities) using four items per domain. Raw scores range from 4 to 20 for each health domain and there are t-scores for each domain. Higher score in physical function, cognitive function, & ability to participate in social roles & activities) indicate good health, and high scores in other domain indicate worse health.
Time Frame: Baseline, 8 weeks, 6 months,12 months
Reporting Status: Not Posted, anticipated posting 2026-05

5. Secondary Outcome: Opioid Prescription Use at Baseline, 8 Weeks, 6 Months, and 12 Months
Description: The Current Opioid Misuse Measure® (COMM) will be used to assess opioid prescription use. It is a 17-item, patient self-assessment measure designed to identify individuals taking opioids. Scoring is based on a Likert 5-point scale from 0 (never) to 4 (very often). A score of 9 or above is a positive indicator, ie, participant has been identified as misusing his/her medication and is at an increased risk of abuse.
Time Frame: Baseline, 8 weeks, 6 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

6. Secondary Outcome: Mindfulness at Baseline, 8 Weeks, 6 Months, & 12 Months
Description: Mindfulness will be assessed by the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), 12-item scale that measures everyday mindfulness and focuses on the degree to which respondents experience their thoughts and feelings. Items are rated on a 4-point Likert scale from 1 (rarely/not at all) to 4 (almost always). Scores on the scale are summed. Higher scores reflect greater mindfulness.
Time Frame: Baseline, 8 weeks, 6 months,12 months
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Mindfulness at 12 Months
Description: Mindfulness will be assessed by the Global Mindfulness Measure at 12 months. Items are rated on a 5-point Likert scale from 1 (rarely/not at all) to 5 (very much). Scores on the scale are summed. Higher scores reflect greater mindfulness.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Patient Impression of Change at 8 Weeks, 6 Months, & 12 Months
Description: Patient impression of change is assessed by the self-report measure Patient Global Impression of Change (PGIC) reflects a respondent's belief about the efficacy of treatment to their pain. This single-item scale is rated on a 6-point Likert scale from 0 (very much improved) to 6 (very much worse).
Time Frame: 8 weeks, 6 months,12 months
Reporting Status: Not Posted, anticipated posting 2026-05

9. Secondary Outcome: Pain Catastrophizing at Baseline, 8 Weeks, 6 Months, & 12 Months
Description: Pain catastrophizing will be assessed by the Pain Catastrophizing Scale short form, a 6-item self-report questionnaire that assesses how catastrophic thinking about low back pain affects respondents. Respondents are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is ranged from 0-24, and the higher score indicates greater pain catastrophizing.
Time Frame: Baseline, 8 weeks, 6 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

10. Secondary Outcome: Tobacco, Alcohol, Prescription Medications, and Other Substance Use at Baseline and 12 Months
Description: The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS-1) Tool consists of a 4-item screening for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). If any item in the TAPS-1 has a response other than "Never" then score this item as positive screening.
Time Frame: Baseline and 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

11. Secondary Outcome: Comorbidity at Baseline
Description: Comorbidity will be assessed by the Charlson Co-Morbidity Index (CCI) with 20 items about different health conditions. Respondents are divided into three groups based on their CCI scores: mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; and severe, with CCI scores ≥5.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-05

12. Secondary Outcome: Treatment Expectation at Baseline
Description: Treatment expectation will be assessed by Treatment Expectancy scale (TEX-Q). The scale consists of 6 items, and each item is rated on a 5-point Likert scale from 1(Not at all) to 5 (Very much). Total raw score is ranged from 6 to 35, and t-score is ranged from 26.1 to 70.8. Higher score indicates higher expectation.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-05

13. Secondary Outcome: Telehealth Usability at Baseline and 8 Weeks
Description: The Telehealth Usability Questionnaire short form (TUQ) will be use to assess respondent's experience with telehealth (interface quality, satisfaction, & future use). The scale consists of 7 item, and each item is rated on a 7-point Likert scale from 0 (Strongly Disagree) to 7 (Strongly Agree). The higher the overall average, the higher the usability of the telehealth system.
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted, anticipated posting 2026-05

14. Secondary Outcome: Anxiety at Baseline
Description: Anxiety will be assessed by the Generalized Anxiety Disorder 2-item (GAD-2), a brief screening tool for generalized anxiety disorder (GAD) and other common anxiety disorders, such as panic disorder, social anxiety disorder, and posttraumatic stress disorder. Each item is ranged from 0 (not at all) to 3 (Nearly every day). The total GAD-2 score ranges from 0-6, and the cut-off point is 3. A score of ≥ 3 on the GAD-2 has been identified as an acceptable cut-off for identifying clinically significant anxiety symptoms in the general population.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-05

15. Secondary Outcome: Depression at Baseline
Description: Depression will be assessed by the Patient Health Questionnaire 2-item (PHQ-2), a brief screening tool for depression. Each item is ranged from 0 (not at all) to 3 (Nearly every day). The PHQ-2 score ranges from 0-6, and the cut-off point is 3. A score of ≥ 3 on the PHQ-2 has been identified as an acceptable cut-off for identifying clinically significant anxiety symptoms in the general population.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-05

16. Secondary Outcome: Sleep Duration at Baseline and 6 Months
Description: Sleep duration will be assessed by a single-item survey asking the amount of actual sleep the respondent got at night per night in the last month in hours and minutes.
Time Frame: Baseline, 6 months
Reporting Status: Not Posted, anticipated posting 2026-05

17. Secondary Outcome: Classes of Back Pain Medication
Description: This outcome will be assessed by the count of participants that take the following pain medication classes: Acetaminophen, NSAIDs (Aspirin, Ibuprofen, Motrin), Muscle Relaxants, Antidepressants, and Opioids
Time Frame: Baseline, 8 weeks, 6 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

18. Secondary Outcome: Amount of Opioid Pain Medication
Description: This outcome will be assessed by determining Morphine Milligram Equivalents (MME) for opioid medications.
Time Frame: Baseline, 8 weeks, 6 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

19. Secondary Outcome: Trauma at 8 Weeks
Description: Trauma will be assessed by the Life Events Checklist (LEC-5) is a self-report measure that assesses exposure to 17 potentially traumatic events in a respondent's lifetime. Respondents indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point nominal scale, and respondents may endorse multiple levels of exposure to the same trauma type. The LEC-5 does not yield a total score or composite score.
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2026-05

20. Secondary Outcome: Chronic Overlapping Pain at 8 Weeks
Description: Chronic overlapping pain will be assessed by the Chronic Overlapping Pain Conditions Screener (COPCs), an assessment tool that helps in the identification of different COPCs that may co-exist within a given individual. The screener consists of 10 COPC conditions and identifies the number of conditions co-occur within a given individual.
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2026-05

21. Secondary Outcome: Dietary Supplement and Natural Products Use at 1 Month
Description: Dietary supplement and natural product use will be assessed by a 10-item questionnaire. The questionnaire identifies if the respondents may have used any dietary supplement and natural products for chronic low back pain management in the past 30 days.
Time Frame: Once at any timepoint
Reporting Status: Not Posted, anticipated posting 2026-05

22. Secondary Outcome: Use of Healthcare Resources by Participants as Documented in the EHR
Description: The electronic health record (EHR) will be reviewed of each participants to ascertain the healthcare resources used.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Adverse events were collected from participants over a 12-month period, which corresponded to the duration of their participation in the study.
Description: Adverse Event: any untoward medical occurrence (whether physical or psychological) associated with the use of meditation or mind and body methods, or breach of confidentiality and which may have a causal relationship with the study procedures.
  This definition is more specific to breach of confidentiality and any issues related to meditation practices.
Arm/Group | Mindfulness Pain Program + Usual PCP Care | Usual PCP Care
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/227
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/227
Other Adverse Events (participants affected / at risk) | 4/224 | 0/227
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Pain Program + Usual PCP Care (N=224) | Usual PCP Care (N=227)
Increased pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The subject reported experiencing increased neck pain, headaches, and nausea, which they attributed to the chair yoga and stretching from a previous session.
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) — The participant felt anxious when lying down regularly.
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — The participant experienced severe nausea during meditation, which also occurred in previous sessions.
Sciatic Pain (Nervous system disorders) | 1 (1) | 0 (0) — The subject stated that they experienced a sciatic flare that began after a meditation session. They complained of pain attributed to the sitting position during the session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04129450/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04129450/ICF_000.pdf